CLINICAL TRIAL: NCT07294261
Title: A Multicenter, Prospective Clinical Study Evaluating Goselasib Combination Therapy for First-Line Treatment of KRAS G12C Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Garsorasib In KRAS G12C Mutant Locally Advanced and Metastatic NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Zhang, MD, Li zhang, DOCTOR SUN YAT-SEN UNVERISITY CANCER CENTER, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-331-01
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Local Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort1: PD-L1≧1%, Garsorasib+Benmelstobart+Anlotinib (Experimental): Histologically confirmed KRAS G12C mutant and PD-L1≧1% local advanced or metastatic NSCLC, at least 1 measurable lesion (RECIST 1.1) ECOG 0-1, treatment naive patients, first step enroll 6-9 patients, 3+3 dose escalation study start with Garsorasib 400mg qd. Patients randomised to Cohort1 or Cohort2. Garsorasib RP2D QD D1-21, Benmelstobart 1200 mg IV D1, q21d, Anlotinib 8mg QD, D1-14,q21d. N1=20 participants.
  Interventions: Drug: Garsorasib, Benmelstobart, Anlotinib
- Cohort2: PD-L1≧1%, Benmelstobart+Anlotinib (Experimental): Histologically confirmed KRAS G12C mutant and PD-L1≧1% local advanced or metastatic NSCLC, at least 1 measurable lesion (RECIST 1.1) ECOG 0-1, treatment naive patients.
  Interventions: Drug: Benmelstobart, Anlotinib
- Cohort3: PD-L1<1%, Garsorasib+Cetuximab Beta Injection (Experimental): Histologically confirmed KRAS G12C mutant and PD-L1<1% local advanced or metastatic NSCLC, at least 1 measurable lesion (RECIST 1.1) ECOG 0-1, treatment naive patients
  Interventions: Drug: Garsorasib, Cetuximab Beta Injection

INTERVENTIONS:
Drug: Garsorasib, Benmelstobart, Anlotinib — Cohort1: Garsorasib RP2D QD D1-21, Benmelstobart 1200 mg IV D1, q21d, Anlotinib 8mg QD, D1-14,q21d. N1=20 participants.
  Arms: Cohort1: PD-L1≧1%, Garsorasib+Benmelstobart+Anlotinib
Drug: Benmelstobart, Anlotinib — Benmelstobart 1200 mg IV D1, q21d, Anlotinib 8mg QD, D1-14,q21d. N2=20 participants.
  Arms: Cohort2: PD-L1≧1%, Benmelstobart+Anlotinib
Drug: Garsorasib, Cetuximab Beta Injection — Garsorasib 600mg BID, D1, q14d, Cetuximab Beta Injection 500mg/㎡ IV, q14d. N3=20 participants
  Arms: Cohort3: PD-L1<1%, Garsorasib+Cetuximab Beta Injection

SUMMARY:
This study is aimed to evaluate the efficacy and safety of the Garsorasib combination therapy in KRAS G12C mutant locally advanced and metastatic NSCLC

ELIGIBILITY:
Inclusion Criteria:

* 1. A written informed consent form should be signed prior to any study-related procedures 2. Male or female, aged 18 or above. 3.Histologically confirmed IIIB-IV NSCLC. 4.Subjects have not received systemic treatment for locally advanced or metastatic non-small cell lung cancer. 5.The patients should be confirmed with KRAS G12C mutation and provide PD-L1 test result. 6.At least 1 measurable lesion (RECIST 1.1 criteria). 7.ECOG 0-1. 8. Good organ function includes:
* Neutrophil count≥1.5×109/L,
* Platelet count≥90×109/L,
* Hemoglobin≥90g/L
* Serum creatinine≤1.5×upper limit of normal (ULN), creatinine clearance≥50 mL/min (Cockcroft-Gault formula)
* Total bilirubin≤1.5×ULN
* AST and ALT≤2.5×ULN; for patients with liver metastasis, AST and ALT≤5×ULN, the investigator should determine whether they are enrolled
* Normal coagulation function: INR and PT≤1.5×ULN ,APTT≤1.5×ULN
* Urinary protein in routine urinalysis is less than 2+, or 24-hour urinary protein quantification is < 1 g.

  9. Life expectancy is at least 3 months; 10.Negative pregnancy test at enrollment. Male or female subjects should commit to take adequate and effective contraceptive measures or abstain from sexual for the duration of study participation and within 3 months after the last dose of the study drug

Exclusion Criteria:

* 1.Patients received anti-tumor drug treatment or investigational drug treatment 3 years ago.2.Non-Small Cell Lung Cancer (NSCLC) with a history of other actionable driver gene mutations for which standard treatment drugs are available (e.g., EGFR, ALK, BRAF(V600E), HER-2, MET(exon14), ROS1, RET, or NTRK1/2/3, etc.) 3.Other active malignant tumors requiring concurrent treatment 4.Patients with active brain metastasis, cancerous meningitis, spinal cord compression, or with brain or pia mater diseases detected by CT or MRI at screening time (patients with stable symptoms and complete treatment 14 days before enrollment may be admitted to the group, but no symptoms of cerebral hemorrhage should be confirmed by craniocerebral MRI, CT or venography evaluation).5.Serious cardiovascular history:
* NYHA (New York Heart Association) Class 3 and 4 congestive heart failure
* Arrhythmia requiring therapeutic intervention
* Thrombotic or embolic event within the past 6 months, e.g., cerebrovascular accident (including transient ischemic attack), and pulmonary embolism
* LVEF<50%
* Subjects with a prolonged QT interval corrected by the Fridericia formula (QTcF) at rest, where the QTcF measured by electrocardiogram (ECG) is > 470 ms in females or > 450 ms in males; or subjects with risk factors for torsades de pointes (TdP), such as hypokalemia deemed clinically significant by the investigator, a family history of long QT syndrome, or a family history of arrhythmias (e.g., pre-excitation syndrome).
* Uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥ 90 mmHg, despite using the optimal medical treatment; 6.Subjects with arterial/venous thrombotic events occurring within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism; or subjects with hypertensive crisis or hypertensive encephalopathy.7.Subjects with a previous history of epilepsy.8.Presence of superior vena cava syndrome.9.Active non-infectious pneumonia with interstitial changes such as interstitial lung disease, radiation pneumonitis, or immune-related pneumonitis during the screening period; active pulmonary tuberculosis; pneumoconiosis; other types of pneumonia graded ≥ Grade 2; or severe impairment of pulmonary function confirmed by pulmonary function tests (FEV1, DLCO, or DLCO/VA < 40% of the predicted value).10.Presence of severe bone damage caused by bone metastases, or a risk of such damage occurring after enrollment-for example, pathological fractures of weight-bearing bones that have occurred within 6 months or may occur after enrollment, extensive bone metastases, or spinal cord compression; or uncontrolled pain related to bone metastases.11.Active or uncontrolled severe infection (≥ CTCAE Grade 2 infection) or unexplained fever > 38.5°C. 12.Third-space fluid accumulation (including pleural effusion, ascites, or pericardial effusion) that is poorly controlled clinically or requires local symptomatic management such as percutaneous drainage. 13.Imaging (CT or MRI) shows that the tumor invades large blood vessels or has an unclear boundary with large blood vessels.14.Subjects with evidence of or a history of bleeding tendency within 2 months prior to the first dose, regardless of severity; subjects with a history of hemoptysis (> 2.5 ml/day) within 2 weeks prior to the first dose, or with unhealed wounds, ulcers, or fractures.15.Known gastrointestinal (GI) dysfunction or gastrointestinal (GI) diseases that may significantly affect the absorption or metabolism of oral medications.16.Have received a live-attenuated preventive vaccine within 4 weeks prior to the first dose.17.Subjects who have experienced severe hypersensitivity reactions after receiving other monoclonal antibody drugs.18.Active autoimmune diseases requiring systemic treatment that occurred within 2 years. 19.Immunodeficiency, or ongoing systemic glucocorticoid treatment, or any other form of immunosuppressive therapy. 20.Active viral infections such as HIV, hepatitis B, hepatitis C, etc. 21.Active syphilis.22.Subjects with renal failure requiring hemodialysis or peritoneal dialysis. 23.Uncontrolled diabetes, FBG>10mmol/L. 24.Received organ transplantation or planned to undergo organ transplantation. 25.Undergone major surgical treatment or significant traumatic injury within 4 weeks. 26.Received palliative radiotherapy for local lesions within 2 weeks. 27.Toxicity of any previous therapy have not recovered to ≤ CTCAE Grade 1 or baseline 28.Pregnant or breeding women. 29.Severe psychiatric or psychological disorders, a history of substance abuse, or a history of severe alcoholism. 30.Allergy to the investigational medicinal product or any of its excipients. 31. The patient is not appropriate for the study In the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 180 days
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).
DoR | up to 180 days
  DoR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
PFS | up to 180 days
  defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
DCR | up to 180 days
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease(SD).
TTR | up to 180 days.
  TTR was defined as Time from Randomization to First Response According to RECIST 1.1 Criteria
OS | up to 360 days.
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yaeger R, Weiss J, Pelster MS, Spira AI, Barve M, Ou SI, Leal TA, Bekaii-Saab TS, Paweletz CP, Heavey GA, Christensen JG, Velastegui K, Kheoh T, Der-Torossian H, Klempner SJ. Adagrasib with or without Cetuximab in Colorectal Cancer with Mutated KRAS G12C. N Engl J Med. 2023 Jan 5;388(1):44-54. doi: 10.1056/NEJMoa2212419. Epub 2022 Dec 21. PMID 36546659
- [Result] Huang L, Guo Z, Wang F, Fu L. KRAS mutation: from undruggable to druggable in cancer. Signal Transduct Target Ther. 2021 Nov 15;6(1):386. doi: 10.1038/s41392-021-00780-4. PMID 34776511
- [Result] Molina-Arcas M, Downward J. Exploiting the therapeutic implications of KRAS inhibition on tumor immunity. Cancer Cell. 2024 Mar 11;42(3):338-357. doi: 10.1016/j.ccell.2024.02.012. PMID 38471457